CLINICAL TRIAL: NCT05794230
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers in India and the Republic of South Africa
Brief Title: Study of a Quadrivalent Meningococcal Conjugate Vaccine (MenACYW Conjugate Vaccine) Given With Routine Pediatric Vaccines in Healthy Infants and Toddlers in India and the Republic of South Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEQ00064; U1111-1225-0926 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Meningococcal Immunisation; Healthy Volunteers
MeSH Terms: interventions — Meningococcal Vaccines; Poliovirus Vaccines; 13-valent pneumococcal vaccine; Measles-Mumps-Rubella Vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; DTaP-IPV-HB-PRP-T vaccine; Hepatitis A Vaccines; Rotavirus Vaccines; RotaTeq; Measles Vaccine

STUDY DESIGN:
Intervention Model Description: Cohort I: Infants and toddlers 6 months to 16 months of age. Eligible participants are randomized in a 1:1 ratio to receive 2 injections of either MenACYW conjugate vaccine (Groups 1 and 3) or Menactra vaccine (Groups 2 and 4), co-administered with routine pediatric vaccines.
  Cohort II: Infants and toddlers 6 weeks to 15 months of age. Eligible participants are randomized in a 2:1 ratio to receive either 3 injections of MenACYW conjugate vaccine co-administered with routine pediatric vaccines (Groups 5 and 7), or routine pediatric vaccines only (Groups 6 and 8).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Groups 1a, 1b and 1c Cohort Ia (India) (Experimental): 2 injections of MenACYW conjugate vaccine: at 6 months of age and second dose at 12 months of age (group 1a) or at 15 months of age (group 1b) or at 16 months of age (group 1c) + co-administered routine pediatric vaccines
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; Biological: Pneumoccocal Vaccine; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: DTwP-HepB-Hib-IPV vaccine; Biological: Hepatitis A vaccine; Biological: Rotavirus vaccine; Biological: Typhoid conjugate vaccine (TCV); Biological: Varicella vaccine live
- Group 2 Cohort Ia (India) (Active Comparator): 2 injections of Menactra vaccine: at 9 months of age and second dose at 16 months of age + co-administered routine pediatric vaccines
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine; Biological: Pneumoccocal Vaccine; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: DTwP-HepB-Hib-IPV vaccine; Biological: Hepatitis A vaccine; Biological: Rotavirus vaccine; Biological: Typhoid conjugate vaccine (TCV); Biological: Varicella vaccine live
- Groups 3 Cohort Ib (RSA) (Experimental): 2 injections of MenACYW conjugate vaccine: at 6 months of age and second dose between 12 and 16 months of age + co-administered routine pediatric vaccines
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; Biological: Oral bivalent types 1 and 3; Poliomyelitis Vaccine (OPV); Biological: Pneumoccocal Vaccine; Biological: DTaP-IPV-Hib-HepB vaccine; Biological: Rotavirus vaccine; Biological: Measles vaccine; Biological: Varicella vaccine live; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: Hepatitis A vaccine
- Group 4 Cohort Ib (RSA) (Active Comparator): 2 injections of Menactra vaccine: at 9 months of age and second dose between 12 and 16 months of age + co-administered routine pediatric vaccines
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine; Biological: Oral bivalent types 1 and 3; Poliomyelitis Vaccine (OPV); Biological: Pneumoccocal Vaccine; Biological: DTaP-IPV-Hib-HepB vaccine; Biological: Rotavirus vaccine; Biological: Measles vaccine; Biological: Varicella vaccine live; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: Hepatitis A vaccine
- Groups 5a and 5b Cohort IIa (India) (Experimental): 3 injections of MenACYW conjugate vaccine: at 6-8 weeks of age and second dose at 14-16 weeks of age with a booster dose administered at 12 months of age (group 5a) or at 15 months of age (group 5b) + co-administered routine pediatric vaccines
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; Biological: Pneumoccocal Vaccine; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: DTwP-HepB-Hib-IPV vaccine; Biological: Hepatitis A vaccine; Biological: Rotavirus vaccine; Biological: Typhoid conjugate vaccine (TCV); Biological: Varicella vaccine live
- Group 6 Cohort IIa (India) (Other): routine pediatric vaccines only
  Interventions: Biological: Pneumoccocal Vaccine; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: DTwP-HepB-Hib-IPV vaccine; Biological: Hepatitis A vaccine; Biological: Rotavirus vaccine; Biological: Typhoid conjugate vaccine (TCV); Biological: Varicella vaccine live
- Group 7 Cohort IIb (RSA) (Experimental): 3 injections of MenACYW conjugate vaccine: at 6-8 weeks of age and second dose at 14-16 weeks of age with a booster dose administered between 12 and 15 months of age + co-administered routine pediatric vaccines
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine; Biological: Oral bivalent types 1 and 3; Poliomyelitis Vaccine (OPV); Biological: Pneumoccocal Vaccine; Biological: DTaP-IPV-Hib-HepB vaccine; Biological: Rotavirus vaccine; Biological: Measles vaccine; Biological: Varicella vaccine live; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: Hepatitis A vaccine
- Group 8 Cohort IIb (RSA) (Other): routine pediatric vaccines only
  Interventions: Biological: Oral bivalent types 1 and 3; Poliomyelitis Vaccine (OPV); Biological: Pneumoccocal Vaccine; Biological: DTaP-IPV-Hib-HepB vaccine; Biological: Rotavirus vaccine; Biological: Measles vaccine; Biological: Varicella vaccine live; Biological: Measles, Mumps, and Rubella Vaccine live (MMR); Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — Liquid solution - intramuscular
  Other Names: MenACYW conjugate vaccine - MenQuadfi™
  Arms: Group 7 Cohort IIb (RSA); Groups 1a, 1b and 1c Cohort Ia (India); Groups 3 Cohort Ib (RSA); Groups 5a and 5b Cohort IIa (India)
Biological: Meningococcal (Groups A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — Liquid solution - intramuscular
  Other Names: Menactra®
  Arms: Group 2 Cohort Ia (India); Group 4 Cohort Ib (RSA)
Biological: Oral bivalent types 1 and 3; Poliomyelitis Vaccine (OPV) — Oral suspension - oral
  Other Names: BIOPOLIO® B1/3
  Arms: Group 4 Cohort Ib (RSA); Group 7 Cohort IIb (RSA); Group 8 Cohort IIb (RSA); Groups 3 Cohort Ib (RSA)
Biological: Pneumoccocal Vaccine — Suspension for injection - intramuscular
  Other Names: Prevnar 13®
Biological: Measles, Mumps, and Rubella Vaccine live (MMR) — Lyophilized powder for injection - subcutaneous
  Other Names: TRESIVAC® PFS
  Arms: Group 2 Cohort Ia (India); Group 6 Cohort IIa (India); Groups 1a, 1b and 1c Cohort Ia (India); Groups 5a and 5b Cohort IIa (India)
Biological: DTwP-HepB-Hib-IPV vaccine — Suspension - intramuscular
  Other Names: EasySix™
  Arms: Group 2 Cohort Ia (India); Group 6 Cohort IIa (India); Groups 1a, 1b and 1c Cohort Ia (India); Groups 5a and 5b Cohort IIa (India)
Biological: DTaP-IPV-Hib-HepB vaccine — Liquid solution - intramuscular
  Other Names: Hexaxim®
  Arms: Group 4 Cohort Ib (RSA); Group 7 Cohort IIb (RSA); Group 8 Cohort IIb (RSA); Groups 3 Cohort Ib (RSA)
Biological: Hepatitis A vaccine — Lyophilized powder for injection - subcutaneous
  Other Names: Biovac®-A
  Arms: Group 2 Cohort Ia (India); Group 6 Cohort IIa (India); Groups 1a, 1b and 1c Cohort Ia (India); Groups 5a and 5b Cohort IIa (India)
Biological: Rotavirus vaccine — Oral solution - oral
  Other Names: RotaTeq®
Biological: Typhoid conjugate vaccine (TCV) — Suspension for injection - intramuscular
  Other Names: Typbar TCV®
  Arms: Group 2 Cohort Ia (India); Group 6 Cohort IIa (India); Groups 1a, 1b and 1c Cohort Ia (India); Groups 5a and 5b Cohort IIa (India)
Biological: Measles vaccine — Freeze-dried powder for reconstitution and injection - subcutaneous
  Other Names: MeasBio®
  Arms: Group 4 Cohort Ib (RSA); Group 7 Cohort IIb (RSA); Group 8 Cohort IIb (RSA); Groups 3 Cohort Ib (RSA)
Biological: Varicella vaccine live — Sterile powder and diluent for injection - subcutaneous
  Other Names: VARIPED®
  Arms: Group 2 Cohort Ia (India); Group 6 Cohort IIa (India); Groups 1a, 1b and 1c Cohort Ia (India); Groups 5a and 5b Cohort IIa (India)
Biological: Varicella vaccine live — Lyophilized powder for injection - subcutaneous
  Other Names: ONVARA®
  Arms: Group 4 Cohort Ib (RSA); Group 7 Cohort IIb (RSA); Group 8 Cohort IIb (RSA); Groups 3 Cohort Ib (RSA)
Biological: Measles, Mumps, and Rubella Vaccine live (MMR) — Lyophilized powder for injection - subcutaneous
  Other Names: OMZYTA®
  Arms: Group 4 Cohort Ib (RSA); Group 7 Cohort IIb (RSA); Group 8 Cohort IIb (RSA); Groups 3 Cohort Ib (RSA)
Biological: Hepatitis A vaccine — Suspension for injection - intramuscular
  Other Names: Avaxim® 80 U Pediatric
  Arms: Group 4 Cohort Ib (RSA); Group 7 Cohort IIb (RSA); Group 8 Cohort IIb (RSA); Groups 3 Cohort Ib (RSA)

SUMMARY:
This open label randomized study will be conducted to evaluate and/or describe the immunogenicity and describe the safety of MenACYW conjugate vaccine when administered in infants and toddlers.

It will be conducted in India and the RSA in 2 cohorts:

* Cohort I: Infants and toddlers 6 months to 16 months of age (Cohort I)
* Cohort II: Infants and toddlers 6 weeks to 15 months of age (Cohort II) In Cohort I, eligible participants will be randomized in a 1:1 ratio to receive 2 intramuscular (IM) injections (1+1 vaccination schedule) of either MenACYW conjugate vaccine (Groups 1 and 3) or Menactra vaccine (Groups 2 and 4), co-administered with routine pediatric vaccines.

In Cohort II, eligible participants will be randomized in a 2:1 ratio to receive either 3 IM injections (2+1 vaccination schedule) of MenACYW conjugate vaccine co-administered with routine pediatric vaccines (Groups 5 and 7) or routine pediatric vaccines only (Groups 6 and 8).

The primary objectives of this study are:

* To demonstrate the non-inferiority of immunogenicity of 2 doses of MenACYW conjugate vaccine compared to 2 doses of Menactra® vaccine in infants and toddlers 6 months to 16 months of age (Cohort I) in terms of serum bactericidal assay using human complement (hSBA) seroprotection (titers ≥ 1:8) in India and the Republic of South Africa (RSA)
* To demonstrate the vaccine immune sufficiency of 3 doses of MenACYW conjugate vaccine in infants and toddlers 6 weeks to 15 months of age (Cohort II) in terms of hSBA seroprotection (titers ≥ 1:8) in India and the RSA

The secondary objectives of this study are:

* To describe the antibody titers to the meningococcal serogroups A, C, Y, and W:

  * before and 30 days post primary series of MenACYW conjugate vaccine and before and 30 days post booster dose of MenACYW conjugate vaccine in infants and toddlers 6 weeks to 15 months of age (Cohort II) in India and the RSA when administered concomitantly with other age-recommended vaccines.
  * before and after 30 days post each dose of MenACYW conjugate vaccine or Menactra vaccine in infants and toddlers 6 months to 16 months of age (Cohort I) in India and the RSA when administered concomitantly with other age-recommended vaccines.
* To describe the antibody responses against the antigens of the other age-recommended vaccines when administered concomitantly with MenACYW conjugate vaccine:

  * in infants and toddlers 6 weeks to 15 months of age (Cohort II) in India and the RSA.
  * in infants and toddlers 6 months to 16 months of age (Cohort I) in India and the RSA.
* To describe the safety profile of MenACYW conjugate vaccine and that of licensed Menactra vaccine in infants and toddlers 6 months to 16 months of age (Cohort I) in India and the RSA when administered concomitantly with other age-recommended vaccines.
* To describe the safety profile of MenACYW conjugate vaccine in infants and toddlers 6 weeks to 15 months of age (Cohort II) in India and the RSA when administered concomitantly with other age-recommended vaccines.
* To describe the safety profile of age-recommended vaccines:

  * in infants 6 weeks to 15 months of age (Cohort II) in India and the RSA when administered concomitantly with MenACYW conjugate vaccine.
  * in infants and toddlers 6 months to 16 months of age (Cohort I) in India and the RSA when administered concomitantly with MenACYW conjugate vaccine.

The duration of each participant's active participation in the study will be approximately 10 to 11 months for Cohort I and 13,5 to 14,5 months for Cohort II.

DETAILED DESCRIPTION:
The duration of each participant's active participation in the study will be approximately 10 to 11 months for Cohort I and 13,5 to 14,5 months for Cohort II.

ELIGIBILITY:
Inclusion Criteria:

* Cohort I: 6 months of age (180 to 209 days of age) on the day of the first study visit
* Cohort II: 6-8 weeks of age (42 to 62 days of age) on the day of the first study visit
* Healthy infants as determined by medical history, physical examination, and judgment of the Investigator
* Participant and parent/ legally acceptable representative (LAR) are able to attend all scheduled visits and to comply with all study procedures
* Cohort I: Z-score ≥ -2 SD on the Weight-for-age table of the WHO Child Growth Standards.
* Cohort II: Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency*; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).

  *Note: Participants with a history of HIV but without evident severe immunosuppression can be included.
* Family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* Individuals with active tuberculosis.
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the study (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* History of intussusception.
* History of any neurologic disorders, including any seizures and progressive neurologic disorders.
* History of Guillain-Barré syndrome (GBS).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the study or to a vaccine containing any of the same substances, including neomycin, gelatin, and yeast.
* Verbal report of thrombocytopenia, as reported by the parent/LAR, contraindicating IM vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination in the Investigator's opinion.
* Chronic illness (including, but not limited to, cardiac disorders, congenital heart disease, chronic lung disease, renal disorders, auto-immune disorders, diabetes, psychomotor diseases, and known congenital or genetic diseases) that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of any vaccine in the 4 weeks preceding the first study vaccination (except for Bacille Calmette-Guérin [BCG], birth dose OPV and birth dose of HepB vaccine) or planned receipt of any vaccine in the 4 weeks following each study vaccination except for the following vaccinations, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines, multivalent influenza vaccines, any COVID-19 vaccines, and administration of OPV on National Immunization Day in India.
* Previous vaccination against meningococcal disease with either the study vaccine or another vaccine (ie, mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup-containing vaccine).
* For Cohort II: Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis (other than birth dose of OPV), Hepatitis A, measles, mumps, rubella, varicella; and of Hib, Streptococcus pneumoniae, and/or RV infection or disease.
* For Cohort II: Previous vaccination with more than 1 dose of HepB vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 6 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1528 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with anti-meningococcal serogroups A, C, Y, W antibody titers above predefined thresholds after 2 doses of MenACYW conjugate vaccine compared to 2 doses of Menactra® vaccine in infants and toddlers 6 months to 16 months of age | 30 days after the second vaccination
  Antibody (Ab) titers against meningococcal serogroups A, C, Y, and W will be measured in infants and toddlers 6 months to 16 months of age ([Group 1 + Group 3] versus [Group 2 + Group 4])
  The following threshold values will be considered: ≥ 1:8
Percentage of participants with anti-meningococcal serogroups A, C, Y, W Ab titers above predefined thresholds after 3 doses of MenACYW conjugate vaccine in infants and toddlers 6 weeks to 15 months of age | 30 days after the booster vaccination
  Ab titers against meningococcal serogroups A, C, Y, and W will be measured in infants and toddlers 6 months to 15 months of age (Group 5 + Group 7)
  The following threshold values will be considered: ≥ 1:8

SECONDARY OUTCOMES:
Geometric Mean Titers (GMTs) of Ab against meningococcal serogroups A, C, Y, and W when MenACYW conjugate vaccine administered concomitantly with other age-recommended vaccine in infants 6 weeks to 15 months of age | Baseline; 30 days after primary series of vaccination; Before and 30 days after booster vaccination
  Ab titers against meningococcal serogroups A, C, Y, and W will be measured Group 5 versus Group 6 in India Group 7 versus Group 8 in RSA Group 5 + Group 7 versus Group 6 + Group 8
Geometric Mean Titers Ratio (GMTR) of Ab against meningococcal serogroups A, C, Y, and W when MenACYW conjugate vaccine administered concomitantly with other age-recommended vaccine in infants 6 weeks to 15 months of age | Baseline; 30 days after primary series of vaccination; Before and 30 days after booster vaccination
  Ab titers against meningococcal serogroups A, C, Y, and W will be measured Group 5 versus Group 6 in India Group 7 versus Group 8 in RSA Group 5 + Group 7 versus Group 6 + Group 8
GMTs of Ab against meningococcal serogroups A, C, Y, and W when MenACYW conjugate vaccine or Menactra vaccine when administered concomitantly with other age-recommended vaccines in infants and toddlers 6 months to 16 months of age | Baseline; Before and 30 days after each vaccination
  Ab titers after vaccination with MenACYW conjugate vaccine or Menetra® will be measured Group 1 versus Group 2 in India Group 3 versus Group 4 in the RSA Group 1 + Group 3 versus Group 2 + Group 4
GMTR of Ab against meningococcal serogroups A, C, Y, and W when MenACYW conjugate vaccine or Menactra vaccine when administered concomitantly with other age-recommended vaccines in infants and toddlers 6 months to 16 months of age | Baseline; Before and 30 days after each vaccination
  Ab titers after vaccination with MenACYW conjugate vaccine or Menetra® will be measured Group 1 versus Group 2 in India Group 3 versus Group 4 in the RSA Group 1 + Group 3 versus Group 2 + Group 4
Percentage of participants with anti-meningococcal serogroups A, C, Y, and W Ab titers met the predefined criteria when MenACYW conjugate vaccine administered concomitantly with other age-recommended vaccine in infants 6 weeks to 15 months of age | Baseline; 30 days after primary series of vaccination; Before and 30 days after booster vaccination
  Ab titers against meningococcal serogroups A, C, Y, and W will be measured
  * hSBA titer ≥ 1:4 and ≥ 1:8
  * hSBA titer ≥ 4-fold rise from pre-vaccination to post-vaccination
  * hSBA vaccine seroresponse
Percentage of participants with anti-meningococcal serogroups A, C, Y, and W Ab titers met the predefined criteria when MenACYW conjugate vaccine administered concomitantly with other age-recommended vaccine in infants and toddlers 6 to 16 months of age | Baseline; Before and 30 days after each vaccination
  Ab titers after vaccination with MenACYW conjugate vaccine or Menetra® will be measured
  * hSBA titer ≥ 1:4 and ≥ 1:8
  * hSBA titer ≥ 4-fold rise from pre-vaccination to post-vaccination
  * hSBA vaccine seroresponse
GMCs of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 weeks to 15 months of age | Baseline
  The following Ab concentrations will be measured:
  - Anti-pertussis Ab concentrations (pertussis toxin [PT], filamentous hemagglutinin [FHA]), fimbriae types 2, 3 [FIM], and pertactin [PRN])
GMCR of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 weeks to 15 months of age | Baseline
  The following Ab concentrations will be measured:
  - Anti-pertussis Ab concentrations (pertussis toxin [PT], filamentous hemagglutinin [FHA], fimbriae types 2, 3 [FIM], and pertactin [PRN])
GMCs/GMTs of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 weeks to 15 months of age | -30 days after:-Dose3 of DTwP-HepB-Hib-IPV/DTaP-IPV-Hib-HepB;-1ry series of PCV13;-measles,mumps & rubella: Dose1 in RSA;Dose2 in India;-1st dose of varicella vaccine -30 days at least after booster dose of PCV13 -Before & 30 days after 1ry series of RV
  The following Ab concentrations/titers will be measured:
  * against the antigens of DTwP-HepB-Hib/DTaP-IPV-Hib-HepB
  * against the antigens of PCV13
  * against the antigens of RV (serum RV immunoglobulin [Ig]A)
  * against the antigens of measles, mumps and rubella
  * against the antigens of varicella vaccine
GMCRs/GMTRs of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 weeks to 15 months of age | -30days after:-1ry series of DTwP-HepB-Hib-IPV/DTaP-IPV-Hib-HepB;-1ry series of PCV13;-measles,mumps & rubella:Dose1 in RSA;Dose2 in India;-1st dose of varicella vaccine -30days at least after booster dose of PCV13 -Before&30 days after 1ry series of RV
  The following Ab concentrations/titers will be measured:
  * against the antigens of DTwP-HepB-Hib-IPV/DTaP-IPV-Hib-HepB
  * against the antigens of PCV13
  * against the antigens of RV (serum RV immunoglobulin [Ig]A)
  * against the antigens of measles, mumps and rubella
  * against the antigens of varicella vaccine
Percentage of participants with Ab concentrations/titers met the predefined criteria in infants and toddlers 6 weeks to 15 months of age | - 30 days after dose 3 of DTwP-HepB-Hib/DTaP-IPV-Hib-HepB - 30 days after primary series of PCV13 and 30 days after the booster dose of PCV13
  The following Ab concentrations/titers will be measured:
  * Anti-tetanus Ab ≥ 0.01 International Units (IU)/milliliter (mL), ≥ 0.1 IU/mL and > 1.0 IU/mL
  * Anti-diphtheria Ab ≥ 0.01 IU/mL, ≥ 0.1 IU/mL and > 1.0 IU/mL
  * Anti-polyribosyl-ribitol phosphate (PRP) Ab ≥ 0.15 micrograms (μg)/mL and ≥ 1.0 μg/mL
  * Pertussis vaccine seroresponse for anti-PT, and anti-PT, anti-FHA, anti-FIM, and anti-PRN
  * Anti-hepatitis B surface antigen (HBsAg) Ab ≥ 10 mIU/mL and ≥ 100 mIU/mL
  * Anti-poliovirus types 1, 2, and 3 Ab titers ≥ 1:8
  * Anti-pneumococcal Ab ≥ 0.35 μg/mL and ≥ 1.0 μg/mL
Percentage of participants with Ab concentrations/titers met the predefined criteria in infants and toddlers 6 weeks to 15 months of age | 30 days after: - Primary series of RV - Dose 1 of measles, mumps and rubella in RSA - Dose 2 of measles, mumps and rubella in India - first dose of varicella vaccine
  The following Ab concentrations/titers will be measured:
  * Anti-RV seroresponse
  * Anti-measles Ab concentrations (serostatus cutoff: 255 mIU/mL)
  * Anti-mumps Ab concentrations (serostatus cutoff: 10 Mumps antibody units/mL)
  * Anti-rubella Ab concentrations (serostatus cutoff: 10 IU/mL)
  * Anti-varicella Ab concentrations (serostatus cutoff: 5gpELISA unit/mL)
GMCs/GMTs of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 months to 16 months of age | 30 days after: - first dose of varicella vaccine - the booster dose of PCV13 - Dose 1 of measles, mumps and rubella in RSA - Dose 2 of measles, mumps and rubella in India - after booster dose of DTwP-HepB-Hib-IPV
  The following Ab concentrations will be measured:
  * against the antigens of varicella
  * against the antigens of PCV13
  * against the antigens of measles, mumps and rubella
  * against the antigens of DTwP-HepB-Hib-IPV
GMCRs/GMTRs of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 months to 16 months of age | 30 days after: - first dose of varicella vaccine - the booster dose of PCV13 - Dose 1 of measles, mumps and rubella in RSA - Dose 2 of measles, mumps and rubella in India - after booster dose of DTwP-HepB-Hib-IPV
  The following Ab concentrations/titers will be measured:
  * against the antigen of varicella
  * against the antigens of PCV13
  * against the antigens of measles, mumps and rubella
  * against the antigens of DTwP-HepB-Hib-IPV
Percentage of participants with Ab concentrations/titers met the predefined criteria in infants and toddlers 6 months to 16 months of age | 30 days after: - the booster dose of PCV13 - Dose 1 of measles, mumps and rubella in RSA - Dose 2 of measles, mumps and rubella in India - first dose of varicella vaccine
  The following Ab concentrations/titers will be measured:
  * anti-pneumococcal Ab concentrations ≥ 0.35 μg/mL and ≥ 1.0 μg/mL
  * anti-measles Ab concentrations (serostatus cutoff: 255 mIU/mL)
  * anti-mumps Ab concentrations (serostatus cutoff: 10 Mumps antibody units/mL)
  * anti-rubella Ab concentrations (serostatus cutoff: 10 IU/mL)
  * anti-varicella Ab concentrations (serostatus cutoff: 5gpELISA unit/mL)
GMCs of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 months to 16 months of age | Pre-booster dose vaccination of DTwP-HepB-Hib-IPV
  The following Ab concentrations will be measured:
  - Anti-pertussis Ab concentrations (pertussis toxin [PT], filamentous hemagglutinin [FHA], fimbriae types 2, 3 [FIM], and pertactin [PRN])
GMCR of Ab against the antigens of age-recommended vaccines in infants and toddlers 6 months to 16 months of age | Pre-booster dose vaccination of DTwP-HepB-Hib-IPV
  The following Ab concentrations will be measured:
  - Anti-pertussis Ab concentrations (pertussis toxin [PT], filamentous hemagglutinin [FHA], fimbriae types 2, 3 [FIM], and pertactin [PRN])
Percentage of participants with Ab concentrations/titers met the predefined criteria in infants and toddlers 6 months to 16 months of age | 30 days after booster dose of DTwP-HepB-Hib-IPV
  The following Ab concentrations/titers will be measured:
  * anti-tetanus Ab concentrations ≥ 0.01 IU/mL, ≥ 0.1 IU/mL and ≥ 1.0 IU/mL
  * anti-diphtheria Ab concentrations ≥ 0.01 IU/mL, and ≥ 0.1 IU/mL
  * anti-PRP Ab concentrations ≥ 0.15 µg)/mL and ≥ 1.0 μg/mL
  * pertussis vaccine seroresponse for anti-PT, anti-FHA, anti-FIM, and anti-PRN
  * anti-HBsAg Ab concentrations ≥ 10 mIU/mL and ≥ 100 mIU/mL
  * anti-poliovirus types 1, 2, and 3 Ab titers ≥ 1:8
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Unsolicited (spontaneously reported) systemic AEs
Percentage of participants reporting solicited injection site and systemic reactions | Within 7 days post-vaccination
  Solicited injection site reactions:
  - tenderness, erythema, swelling
  Solicited systemic reactions:
  - fever, vomiting, crying abnormal, drowsiness, appetite lost, irritability
Number of participants reporting unsolicited AEs | Up to Day 31 post-vaccination
  Unsolicited AEs
Number of participants reporting serious adverse events (SAEs) | From Day 1 to Month 18
  SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (15):
- India (10):
  - Investigational Site Number : 3560006, Chennai
  - Investigational Site Number : 3560007, Hyderabad
  - Investigational Site Number : 3560016, Kanpur
  - Investigational Site Number : 3560009, Kolkata
  - Investigational Site Number : 3560011, Manipal
  - Investigational Site Number : 3560013, Mysore
  - Investigational Site Number : 3560004, Mysore
  - Investigational Site Number : 3560003, New Delhi
  - Investigational Site Number : 3560002, Pune
  - Investigational Site Number : 3560001, Pune
- South Africa (5):
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100003, Cape Town
  - Investigational Site Number : 7100006, George
  - Investigational Site Number : 7100005, Johannesburg
  - Investigational Site Number : 7100001, Middelburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: MEQ00064 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25308&tenant=MT_SNY_9011